CLINICAL TRIAL: NCT05474560
Title: Allopurinol Versus Febuxostat: A New Approach for Management of Hepatic Steatosis in Metabolic-Associated Fatty Liver Disease
Brief Title: Febuxostat Versus Allopurinol on Hepatic Steatosis in MAFLD Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Febuxostat versus allopurinol
Record Dates: First submitted 2022-07-13; First posted 2022-07-26 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-02

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Hyperuricemia
Keywords: Fatty liver disease; Hyperuricemia; Allopurinol; Febuxostat
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Hyperuricemia | interventions — Allopurinol; Febuxostat

STUDY DESIGN:
Intervention Model Description: A total of 90 subjects are enrolled in this study. After the initial screening, the subjects were randomly divided into the control group and the drug treatment group. The control group was given lifestyle intervention for 24 weeks, and the experimental group was given febuxostat oral therapy or allopurinol oral therapy on the basis of lifestyle intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Allopurinol group (Experimental): Allopurinol (100 mg/day) plus lifestyle intervention
  Interventions: Drug: Allopurinol (100 mg/day) plus lifestyle intervention
- Febuxostat group (Experimental): Febuxostat (40 mg/day) plus lifestyle intervention
  Interventions: Drug: Febuxostat 40 mg plus lifestyle intervention
- lifestyle intervention (Active Comparator): diet and exercise
  Interventions: Behavioral: Life style intervention

INTERVENTIONS:
Drug: Allopurinol (100 mg/day) plus lifestyle intervention — participants accept allopurinol treatment (100 mg, once a day, orally). Behavioral: lifestyle intervention According to NAFLD guidelines, participants receive lifestyle intervention (diet and exercise).
  Other Names: Allopurinol group
  Arms: Allopurinol group
Drug: Febuxostat 40 mg plus lifestyle intervention — participants accept Febuxostat treatment (100 mg, once a day, orally). Behavioral: lifestyle intervention According to NAFLD guidelines, participants receive lifestyle intervention (diet and exercise).
  Other Names: Febuxostat group
  Arms: Febuxostat group
Behavioral: Life style intervention — According to NAFLD guidelines, participants receive lifestyle intervention (diet and exercise).
  Arms: lifestyle intervention

SUMMARY:
Metabolic associated fatty liver disease (MAFLD) is the most common and harmful chronic liver disease, and it is increasingly diagnosed in many developed and developing countries.

Previous studies suggested a significant association between hyperuricemia and MAFLD and that hyperuricemia plays a causal role in the development of MAFLD.

Xanthine oxidase is a key enzyme in uric acid metabolism, and It thus can be considered as is a therapeutic target for MAFLD, so long-term urate-lowering therapy may play a role in amelioration of MAFLD by controlling uric acid levels. So, this study is conducted to assess the effect of controlling hyperuricemia using different xanthine oxidase inhibitors on amelioration of MAFLD.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effect of urate lowering therapy on improvement of steatosis in metabolic associated fatty liver disease (MAFLD) patients with hyperuricemia, by comparing two xanthine oxidase inhibitors allopurinol (100 mg/day), versus Febuxostat (40 mg/day), versus lifestyle intervention.

Primary Outcome: Regression of hepatic steatosis. Secondary Outcome: Improvement of Serum uric acid and incidence of hepatotoxicity.

Study design: This study is a prospective, interventional three arm study. Setting: Patients will be recruited from the National Hepatology and Tropical Medicine Research institute, Cairo, Egypt.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-65.
* Males and Females
* Metabolic syndrome according to the NCEP ATP III definition [13]: present of three or more of the following five criteria are met:

  * Waist circumference over 40 inches (men) or 35 inches (women), Central obesity - defined as waist circumference ≥ 102 cm for Men and ≥ 88 cm for women
  * Blood pressure over 130/85 mmHg,
  * Basting triglyceride (TG) level over 150 mg/dl,
  * Fasting high-density lipoprotein (HDL) cholesterol level less than 40 mg/dl (men) or 50 mg/dl (women),
  * Fasting blood sugar over 100 mg/dl.
* Serum uric acid levels of > 420μmol/L (>7 mg/dL) in men and >360 μmol/L (>6 mg/dL) women.

Exclusion Criteria:

* Renal insufficiency defined by serum creatinine > 2.0 mg/dl.

  * Patients with obvious abnormal liver function: serum transaminase (ALT, AST, one of them) exceed 2 times the upper limit of normal reference value.
  * Have a history of viral hepatitis, or serological examination suggests hepatitis virus infection, or have a history of other liver diseases.
  * Complementation with diabetes, or fasting blood glucose >7.8mmol/L, or HbA1c >7.5%.
  * Severe hypertension, blood pressure ≥ 160/100 mmHg.
  * A history of allergy to febuxostat and allopurinol; in the acute active phase of gout.
  * Drinking equivalent to alcohol intake ≥30g/d(male), ≥20g/d(female).
  * Complicated coronary heart disease.
  * Cardiac dysfunction (cardiac function grade 2 or above).
  * Patients with asthma and other respiratory diseases.
  * Intestinal diseases such as inflammatory bowel disease.
  * Any history of systemic malignancy in the past 5 years.
  * Use of uric-lowering drugs in the 4 weeks before screening: febuxostat, allopurinol, benzbromarone.
  * Morbid obesity (BMI>37.5kg/m2).
  * Triglyceride ≥5.0 mmol/L was found to be significantly abnormal in baseline examination.
  * had received systemic hormone or immunosuppressive therapy within 3 months prior to screening or expected to receive hormone or immunosuppressive therapy in the future.
  * Use of other drugs affecting uric acid metabolism were adjusted within 4 weeks before screening: losartan, fenofibrate, irbesartan, thiazide diuretics, loop medullar diuretics, compound antihypertensive agents containing diuretics.

Other drugs that may affect liver fat content were taken within 4 weeks before screening.

* Women who are lactating or pregnant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-28 (Actual); Study Completion 2023-01-28 (Actual)

PRIMARY OUTCOMES:
Change in hepatic steatosis . | 3 months
  FibroScan instrument measures fibrosis (scarring) and steatosis (fatty changes) in your liver. Fatty changes are when fat builds up in your liver cells.
  FibroScan steatosis result (CAP score): decibels per meter(dB/M). it ranges from 100 to 400 dB/m. The fibrosis result is measured in kilopascals (kpa). It is normaly between 2 and 6 kpa.

SECONDARY OUTCOMES:
Serum uric acid. | three months
  change in serum uric milligrams/deciliter (mg/dl) in hyperuricemia patients. Normal values are 1.5 to 6.0 (mg/dl).

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Ma Zaki, Ass.Prof., Study Director — Ain Shams University
Locations (1):
- National Hepatology and tropical medicine research institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu Z, Que S, Zhou L, Zheng S. Dose-response Relationship of Serum Uric Acid with Metabolic Syndrome and Non-alcoholic Fatty Liver Disease Incidence: A Meta-analysis of Prospective Studies. Sci Rep. 2015 Sep 23;5:14325. doi: 10.1038/srep14325. PMID 26395162
- [Background] Younossi Z, Anstee QM, Marietti M, Hardy T, Henry L, Eslam M, George J, Bugianesi E. Global burden of NAFLD and NASH: trends, predictions, risk factors and prevention. Nat Rev Gastroenterol Hepatol. 2018 Jan;15(1):11-20. doi: 10.1038/nrgastro.2017.109. Epub 2017 Sep 20. PMID 28930295
- [Background] Darmawan G, Hamijoyo L, Hasan I. Association between Serum Uric Acid and Non-Alcoholic Fatty Liver Disease: A Meta-Analysis. Acta Med Indones. 2017 Apr;49(2):136-147. PMID 28790228
- [Background] Allen AM, Therneau TM, Larson JJ, Coward A, Somers VK, Kamath PS. Nonalcoholic fatty liver disease incidence and impact on metabolic burden and death: A 20 year-community study. Hepatology. 2018 May;67(5):1726-1736. doi: 10.1002/hep.29546. Epub 2018 Mar 23. PMID 28941364
- [Background] Turnheim K, Krivanek P, Oberbauer R. Pharmacokinetics and pharmacodynamics of allopurinol in elderly and young subjects. Br J Clin Pharmacol. 1999 Oct;48(4):501-9. doi: 10.1046/j.1365-2125.1999.00041.x. PMID 10583019
- [Background] Lee JS, Won J, Kwon OC, Lee SS, Oh JS, Kim YG, Lee CK, Yoo B, Hong S. Hepatic Safety of Febuxostat Compared with Allopurinol in Gout Patients with Fatty Liver Disease. J Rheumatol. 2019 May;46(5):527-531. doi: 10.3899/jrheum.180761. Epub 2018 Nov 15. PMID 30442825
- [Background] Moy FM, Bulgiba A. The modified NCEP ATP III criteria maybe better than the IDF criteria in diagnosing Metabolic Syndrome among Malays in Kuala Lumpur. BMC Public Health. 2010 Nov 6;10:678. doi: 10.1186/1471-2458-10-678. PMID 21054885
- [Background] Kuo CF, Yu KH, Luo SF, Chiu CT, Ko YS, Hwang JS, Tseng WY, Chang HC, Chen HW, See LC. Gout and risk of non-alcoholic fatty liver disease. Scand J Rheumatol. 2010 Nov;39(6):466-71. doi: 10.3109/03009741003742797. Epub 2010 Jun 21. PMID 20560813
- [Background] Hallsworth K, Adams LA. Lifestyle modification in NAFLD/NASH: Facts and figures. JHEP Rep. 2019 Nov 5;1(6):468-479. doi: 10.1016/j.jhepr.2019.10.008. eCollection 2019 Dec. PMID 32039399
- [Background] Harrison SA, Day CP. Benefits of lifestyle modification in NAFLD. Gut. 2007 Dec;56(12):1760-9. doi: 10.1136/gut.2006.112094. Epub 2007 Oct 2. No abstract available. PMID 17911352